CLINICAL TRIAL: NCT03867838
Title: Effects of Post-Stroke Upper Extremity Assistance
Brief Title: Effects of a Compliant Arm Support on Post-stroke Upper Extremity Range of Motion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Allison Okamura, Professor of Mechanical Engineering, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB-49194; SNI-BI1-02 (Other Grant/Funding Number: Stanford Neurosciences Institute)
Record Dates: First submitted 2019-03-05; First posted 2019-03-08 (Actual); Results first posted 2021-02-23 (Actual); Last update posted 2021-02-23 (Actual); Status verified 2021-02

CONDITIONS: Arm Weakness as a Consequence of Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Stroke survivors (Experimental): Stroke survivors with upper extremity motor impairments
  Interventions: Device: compliant support

INTERVENTIONS:
Device: compliant support — Participants will be given compliant arm support and their reachable workspace measured

SUMMARY:
The aim of this study is to show that a wearable compliant arm support consisting of inflatable bladders with adjustable straps to connect them to the waist and arm can meaningfully increase the reachable workspace of persons with post-stroke arm weakness.

ELIGIBILITY:
Inclusion Criteria:

* greater than 6 months post-stroke
* passive abduction to 90 degrees at shoulder
* reduced active (retro)flexion/extension at shoulder when abducted to 90 degrees
* reduced active flexion/extension at elbow

Exclusion Criteria:

* unable to give informed consent
* unable to comprehend and follow instructions
* have a condition (other than stroke) affecting sensorimotor function
* show evidence of unilateral spatial neglect
* unable to sit in a chair without armrests for 2 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2019-06-14 (Actual); Primary Completion 2020-04-27 (Actual); Study Completion 2020-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Allison Okamura, Principal Investigator — Stanford University
Locations (1):
- Stanford University CHARM Lab, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Simpson CS, Okamura AM, and Hawkes EW. Exomuscle: An inflatable device for shoulder abduction support. 2017 IEEE International Conference on Robotics and Automation (ICRA) 2017; pp. 6651-6657.
- [Result] Simpson C, Huerta B, Sketch S, Lansberg M, Hawkes E, and Okamura A. Upper Extremity Exomuscle for Shoulder Abduction Support. IEEE Transactions on Medical Robotics and Bionics. 2020; 2(3):474-484.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were screened to include only those whose most recent stroke occurred more than 6 months before the study date and to exclude those with conflating health problems, sensory deficits, or that experience pain during passive movements of the arm.
Groups:
- All Participants: Stroke survivors with upper extremity motor impairments
Period: Overall Study
Arm/Group | All Participants
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Participants
Number analyzed (Participants) | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 51 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 4
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Fugl-Meyer Assessment of sensorimotor function [Mean (Standard Deviation); unit: units on a scale] — The Fugl-Meyer Assessment of sensorimotor function is an index for assessing sensory and motor ability after a stroke. Our study considered only the upper extremity portion of this index. This index consists of a series of tasks that are individually assessed by the experimenter on a scale from 0 to 2 where 0 indicates inability to perform the task and 2 indicates faultless execution. The scores of these tasks are summed with a minimum score of 0 indicating severe sensorimotor impairments and a maximum score of 66 indicating no observable sensorimotor impairments.
  units on a scale | 27 (13)
Correct scapulohumeral rhythm [Count of Participants; unit: Participants] — To reduce the risks of adverse events during experimentation, participants were screened by the experimenter for correct scapulohumeral rhythm. Participants were asked to flex the shoulder from 0˚ (arm by the side) to 90˚ (arm parallel to the floor) while the experimenter examined the motion of the scapula. Participants were classified as having correct scapulohumeral rhythm if the scapula began to rotate with shoulder flexion above approximately 30˚ as is typical in people with no sensorimotor impairments.
  Participants | 6
Spatial neglect [Count of Participants; unit: Participants] — Some stroke survivors experience an unawareness of portions of space, a phenomenon called spatial neglect. Spatial neglect was tested clinically by wiggling fingers for two seconds in one or both visual fields (six trials). Neglect was considered to be present when a participant failed at least once to accurately identify the stimulus.
  Participants | 0
Reachable workspace [Mean (Standard Deviation); unit: m^2] — Participants were instructed to individually flex and extend the elbow and shoulder to trace the largest possible circle that they could reach while keeping the hand and elbow raised to the height of the shoulder while the motion of the arm was tracked with motion capture. This protocol was originally developed by Sukal et al., 2007; PubMed ID: 17634933 to asses post-stroke motor abilities. A larger workspace area indicates fewer upper extremity motor impairments.
  m^2 | 0.10 (0.11)
Biceps activation [Mean (Standard Deviation); unit: mV] — Activity in the biceps muscle can become erroneously coupled with activity in the deltoid muscles after a stroke, limiting motor abilities. More information can be found in Beer et al., 2017, PubMed ID: 17486581. To assess the extent of such coupling, we replicated the experiment developed by Ellis et al., 2017, PubMed ID: 28558314, in which the activity of the biceps muscle is measured with surface electromyography while the arm is placed in a posture that activates the deltoid muscle. Larger values of activity indicate more coupling, which may correlate with motor impairment.
  mV | 0.19 (0.25)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Reachable Workspace
Description: Reachable workspace was measured using a PhaseSpace motion capture system, recorded as an area (in square meters).
Time Frame: baseline, while using support device, and 30 minutes following removal of support device (up to 4 minutes per assessment)
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | All Participants
Number analyzed (Participants) | 6
percent change
  On support device | 27 (84)
  Post support device | -71 (41)

2. Secondary Outcome: Percent Change From Baseline in Biceps Activation
Description: Biceps activation measured using surface electromyography during an isometric hold to approximate the contributions of erroneous flexor synergies.
Time Frame: baseline and while using support device (up to 10 seconds per assessment)
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | All Participants
Number analyzed (Participants) | 6
percent change | -16 (71)

ADVERSE EVENTS:
Time Frame: Up to 3 days
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2021-01-08): https://cdn.clinicaltrials.gov/large-docs/38/NCT03867838/Prot_001.pdf